CLINICAL TRIAL: NCT05123352
Title: Investigation of the Gut Microbiota Evaluated by Metagenomic Next-Generation Sequencing (mNGS) in Acute Myeloid Leukemia Receiving Standard Intensive Chemotherapy or Bcl-2 Inhibitor-based Targeted Induction Therapy
Brief Title: Investigation of the Gut Microbiota in Acute Myeloid Leukemia Receiving Two Different Induction Therapies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: AML-GutMicrobiota01
Record Dates: First submitted 2021-10-26; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-10

CONDITIONS: Acute Myeloid Leukemia; Adult; Gut Microbiota; Infections
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard intensive chemotherapy: Patients with acute myeloid leukemia in this cohort will receive standard induction chemotherapy that combines seven days of cytarabine and three days of anthracycline (7+3 regimen).
  Interventions: Other: collection of biological samples and clinical data
- Bcl-2 inhibitor-based targeted therapy: Patients with acute myeloid leukemia in this cohort will receive Bcl-2 inhibitor-based targeted therapy, such as combination of bcl-2 inhibitor plus decitabine/azacitidine with or without sorafenib.
  Interventions: Other: collection of biological samples and clinical data

INTERVENTIONS:
Other: collection of biological samples and clinical data — blood and feces samples

SUMMARY:
In this observational single-center cohort study, metagenomic Next-Generation Sequencing (mNGS) will be used to investigate the features and changes of gut microbiota in acute myeloid leukemia (AML) patients during the treatment of two different induction therapy regimens [standard intensive chemotherapy (7+3) or bcl-2 inhibitor-based targeted therapy].

DETAILED DESCRIPTION:
Infections remain one of the major complications during induction therapy of acute myelocytic leukemia (AML). Previous studies have shown that the variation of gut microbiota was an effective predictor for infection development of AML during induction therapy. A growing number of patients with AML received bcl-2 inhibitor-based targeted induction therapy. The investigators assume that there are different effects of bcl-2 inhibitor-based induction therapy on gut microbiota compared with standard intensive chemotherapy (7+3 regimen). Metagenomic Next-Generation Sequencing (mNGS) will be used to perform the investigation of gut microbiota in AML receiving two different induction therapies. And the relationships of gut microbiota with infection complication will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 65> =Age (years) >= 18;
2. Newly diagnosed as AML patients according to World Health Organization (WHO) classification;
3. Eastern Cooperative Oncology Group (ECOG) Performance status of 0,1,2;
4. Patients will receive standard intensive chemotherapy (7+3) or bcl-2 inhibitor-based targeted therapy;
5. Patients have not received prior therapy for AML (except hydroxycarbamide);
6. Liver function: Total bilirubin lower than 3 upper limit of normal (ULN); Aspartate aminotransferase (AST) lower than 3 ULN; Alanine aminotransferase (ALT) lower than 3 ULN (except extramedullary infiltration of leukemia);
7. Renal function with creatinine clearance rate (Ccr) higher than 30 ml/min;
8. Patients who sign the informed consent must have the ability to understand and be willing to participate in the study and sign the informed consent.

Exclusion Criteria:

1. Acute promyeloid leukemia;
2. AML with central nervous system (CNS) infiltration;
3. Any history of chronic intestinal affections (Crohn disease, inflammatory bowel disease, gluten intolerance) or gastrointestinal surgery;
4. HIV infection, Chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment;
5. Severe and active infection that is difficult to control and cannot tolerate induction therapy;
6. Female who are pregnant, breast feeding or childbearing potential without a negative urine pregnancy test at screen;
7. Antibiotic exposure within 30 days before enrollment (carbapenems and/or tigecycline were not included, penicillin, cephalosporins and quinolones could be included)
8. Patients reject to participate in the study;
9. Patients with severe heart failure (grade 3-4) or patients deemed unsuitable for enrolment by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Candidates will come from patients with newly diagnosed acute myeloid leukemia (AML) in the First Affiliated Hospital of Soochow University from November 2021. Participants should meet the inclusion criteria and not meet exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Changes in gut microbiota composition in patients with acute myeloid leukemia before, during and after induction therapy | Day 0 i.e.: feces sampling is done at time of diagnosis before induction therapy
  Sequencing DNA extracts from patients' feces to obtain the description of gut microbiota composition in those patients
Changes in metabolites composition of blood in patients with acute myeloid leukemia before, during and after induction therapy | Day 0 i.e.: blood sampling is done at time of diagnosis before induction therapy
  Metabolomics performed on patients' blood to report the metabolites composition in those patients

SECONDARY OUTCOMES:
Changes in immune cells of blood in patients with acute myeloid leukemia before, during and after induction therapy | Day 0 i.e.: blood sampling is done at time of diagnosis before induction therapy
  Immunomicin performed on patients' blood to report the composition of immune cells in those patients
Changes of gut permeability markers and microbial compounds of blood in patients with acute myeloid leukemia before, during and after induction therapy | Day 0 i.e.: blood sampling is done at time of diagnosis before induction therapy
  ELISA (in pg/ml)
Infection rate during induction therapy | From date of first one cycle induction therapy start to the end of Cycle 1 (each cycle is 28 days) or death from any cause during Cycle 1 induction therapy.
  Infection rate of patients with acute myeloid leukemia after two different induction therapy
Rate of complete remission | From date of first one cycle induction therapy start to the end of Cycle 1 (each cycle is 28 days) or death from any cause during Cycle 1 induction therapy.
  Complete remission after one cycle of induction therapy
Changes in number of participants with treatment related-related adverse events as assessed by CTCAE v4.0 | From date of first one cycle induction therapy start to the end of Cycle 1 (each cycle is 28 days) or death from any cause during Cycle 1 induction therapy.
  CTCAE (common terminology criteria for adverse event version 4)

CONTACTS AND LOCATIONS:
Overall Officials: Suning Chen, professor, Principal Investigator — The First Affiliated Hospital of Soochow University, Jiangsu Institute of Hematology
Locations (1):
- The First Affiliated Hospital of Soochow University, Jiangsu Institute of Hematology, Suzhou, Jiangsu, China